CLINICAL TRIAL: NCT03186963
Title: Effectiveness of Immobilization in the Postoperative Analgesia of Patients With Distal Radius Fracture Treated With Volar Locking Plating: a Prospective, Randomized Clinical Trial
Brief Title: Effectiveness of Immobilization in the Postoperative Analgesia of Surgically Treated Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernando B Andrade-Silva, MD, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Distalradius
Record Dates: First submitted 2017-01-19; First posted 2017-06-14 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Radius Fracture Distal
Keywords: distal radius fracture; volar plate; immobilization
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No immobilization (Experimental): Patients receive a conventional dressing made with gauze, cotton padding and inelastic bandage after the surgery. They are instructed to start light wrist movements on the first postoperative day and progress as tolerated, beginning rehabilitation with physiotherapy after 2 weeks postoperatively.
  Interventions: Procedure: No immobilization
- Volar splint (Active Comparator): Patients receive a volar plaster splint with inelastic bandage after the surgery, and are instructed not to remove the immobilization for 2 weeks. After this period, the immobilization is removed and patients begin rehabilitation with physiotherapy.
  Interventions: Procedure: Volar splint

INTERVENTIONS:
Procedure: No immobilization — Conventional wrist dressing
  Arms: No immobilization
Procedure: Volar splint — Volar plaster splint
  Arms: Volar splint

SUMMARY:
The purpose of this study is to determine wether postoperative immobilization is effective in controlling the pain of patients with intra-articular distal radius fractures treated with volar locking plate fixation. The study hypotheses is that postoperative immobilization does not enhance the analgesia of these patients.

DETAILED DESCRIPTION:
Volar locking plate fixation has been used as the gold standard treatment for intra-articular distal radius fractures. The need for postoperative immobilization after this type of fixation is controversial, with some authors advocating its use for analgesia. Conversely, the use of immobilization might retard the recovery of wrist range of motion and function. The objective of this study is to compare the level of pain and function of patients undergoing surgical fixation of distal radius fractures using or not postoperative immobilization. Patients will be randomly assigned to receive a plaster splint or conventional dressing immediately after the surgery. The main outcome is the level of pain in the first two weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Intra-articular distal radius fracture treated with volar locking plate fixation;
* Fracture occurred within the prior 30 days;
* Consent to participate in the study

Exclusion Criteria:

* Concomitant fracture of the ipsilateral upper limb
* Previous lesion of the ipsilateral upper limb with functional deficit
* Bilateral fracture
* Concomitant neurologic injury
* Patient not amenable to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-05; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Level of pain | 12 hours
  Visual analogue scale for pain
Level of pain | 18 hours
  Visual analogue scale for pain
Level of pain | 24 hours
  Visual analogue scale for pain
Level of pain | Once a day in the first week
  Visual analogue scale for pain
Level of pain | 2 weeks
  Visual analogue scale for pain

SECONDARY OUTCOMES:
Level of pain | 6 weeks
  Visual analogue scale for pain
Level of pain | 3 months
  Visual analogue scale for pain
Level of pain | 6 months
  Visual analogue scale for pain
DASH score | 6 weeks
  Disabilities of the Arm, Shoulder and Hand (DASH)
DASH score | 3 months
  Disabilities of the Arm, Shoulder and Hand (DASH)
DASH score | 6 months
  Disabilities of the Arm, Shoulder and Hand (DASH)
Wrist flexion-extension arc | 2 weeks
  Assessed by goniometry
Wrist flexion-extension arc | 6 weeks
  Assessed by goniometry
Wrist flexion-extension arc | 3 months
  Assessed by goniometry
Wrist flexion-extension arc | 6 months
  Assessed by goniometry
Forearm rotation arc | 2 weeks
  Assessed by goniometry
Forearm rotation arc | 6 weeks
  Assessed by goniometry
Forearm rotation arc | 3 months
  Assessed by goniometry
Forearm rotation arc | 6 months
  Assessed by goniometry
Tramadol use | Once a day in the first week post-op
  Percentage of patients requesting additional analgesia with tramadol in the first week
Complication | up to 24 weeks
  Percentage of patients presenting with any type of local orthopedic complication

CONTACTS AND LOCATIONS:
Overall Officials: Kodi E Kojima, MD, Study Chair — Institute of Orthopedics - University of Sao Paulo
Locations (1):
- Institute of Orthopedics and Traumatology - University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No